CLINICAL TRIAL: NCT02848482
Title: Anti-infective Effect of Non-surgical Treatment With and Without Photodynamic
Brief Title: Anti-infective Effect of Non-surgical Treatment With and Without Photodynamic Therapy on Initial Peri-implantitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1036_2016
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Peri-implantitis
Keywords: Photodynamic therapy
MeSH Terms: conditions — Peri-Implantitis | interventions — Photochemotherapy; Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Plastic curette will be used to perform the mechanical debridement. Then, irrigation (2% chlorhexidine) will be performed at contaminated sites.
  Interventions: Procedure: Mechanical debridement; Drug: Irrigation
- Test group (Experimental): Plastic curette will be used to perform the mechanical debridement. Then, the addition photodynamic therapy (PDT) will be performed. This will be performed with a set-up for PDT (HELBO Photodynamic Systems, German).
  Interventions: Device: Photodynamic therapy; Procedure: Mechanical debridement

INTERVENTIONS:
Device: Photodynamic therapy — Photodynamic therapy (HELBO Photodynaimc Systems GmbH, Wels, Austria)
  Arms: Test group
Procedure: Mechanical debridement — Plastic scalers (Have implantrecallset, Kerr, Italy) will be used to curette the contaminated sites.
Drug: Irrigation — 0.2% chlorhexidine digluconate solution (Bioworld, Madision, US) will be irrigated at contaminated sites for 1 minute.
  Arms: Control group

SUMMARY:
Photodynamic therapy (PDT), also known as photoradiation therapy, phototherapy, or photochemotherapy, involves the use of a photoactive dye (photosensitizer) that is activated by exposure to light of a specific wavelength in the presence of oxygen. In recent years, PDT has been introduced as an important novel disinfection therapy in the field of implant dentistry. The inactivation of microorganisms using PDT has been defined as antimicrobial PDT. PDT has the potential to be an alternative of antibiotics, especially for the treatment of localized infections and oral biofilm. PDT is unlikely to cause bacterial-resistance and is equally effective against antibiotic-resistance and antibiotic-susceptible bacteria.

Inconsistent results have been reported regarding the potential role of PDT as an adjunct to mechanical debridement in the management of peri-implant infection. Thus, the aim of the present trial is to investigate the treatment effect of non-surgical treatment with and without photodynamic therapy on initial peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages over 18.
2. Subjects with at least one implant with initial peri-implantitis: PPD of 4-6mm combined with BOP+, bone loss of 0.5-2mm on peri-apical radiographs compared to the time point of restoration placement.
3. Availability for the 12 month duration of the study.
4. Good general health (ASA classification I-II).
5. Signed Informed Consent Form.

Exclusion Criteria:

1. Medically compromised subjects (ASA classification III-V)
2. Pregnant or lactating females.
3. Peri-implant mucositis defined as the absence of radiographic marginal bone loss between restoration placement and pre-screening review.
4. Subjects treated for >2 weeks with any medication known to affect soft tissue condition (e.g. phenytoin, calcium antagonists, cyclosporin, Coumadin and non-steroidal anti-inflammatory drugs) within 1 month of the baseline examination.
5. Unwilling to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change of percentage of bleeding on probing sites | From baseline to 12 months after treatment
  A PQW Williams probe (Hu-Friedy, Chicago Ill, USA)will be used to detect the peri-implant pocket. the percentage of bleeding on probing sites (BOP) will be recorded.

SECONDARY OUTCOMES:
Change of Probing Pocket Depth | From baseline to 12 months after treatment
  Probing Pocket Depth at every site will be assessed as the distance from the gingival margin to the apical end of the pocket using a PQW Williams probe (Hu-Friedy, Chicago Ill, USA).
Change of modified plaque index | From baseline to 12 months after treatment
  Modified plaque index 0= No detection of plaque.
  1. Plaque only recognized by running a probe across the smooth marginal surface of the implant. Implants covered by titanium spray in this area always score 1.
  2. Plaque can be seen by the naked eye.
  3. Abundance of soft matter.
Change of clinical attachment level | From baseline to 12 months after treatment
Marginal bone loss | From baseline to 12 months after treatment
  Periapical radiographs will be taken at baseline, 3, 6, 9 and 12 month examination. The distance from implant shoulder to the most coronal level of implant-bone contact at the mesial and distal site will be recorded. The alteration of the distance between baseline and follow-up visit will be defined as marginal bone loss.
Mucosa recession | From baseline to 12 months after treatment
  The distance from mucosa margin to the implant shoulder will be recorded using a PQW Williams probe (Hu-Friedy, Chicago Ill, USA). The alteration of the distance between baseline and follow-up visit will be defined as the mucosa recession.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China